CLINICAL TRIAL: NCT02459301
Title: A Dose-Ranging Study of IPH2201 in Patients With Gynecologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I221
Record Dates: First submitted 2015-05-19; First posted 2015-06-02 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPH2201 (Experimental): Part 1: 1, 4 or 10mg/kg, IV, 1 hour duration on Day 1 every 2 weeks.
  Part 2: Patients will receive single agent IPH2201 as above with the actual dose dependent on the outcome of Part 1
  Interventions: Drug: IPH2201

INTERVENTIONS:
Drug: IPH2201

SUMMARY:
The purpose of this study is to test the safety of a new drug, IPH2201, to see what effects it has on this type of cancer.

DETAILED DESCRIPTION:
This research is being done because there is no treatment that will cure this type of cancer. Although some types of chemotherapy may cause this cancer to shrink for a time, better options are needed. In laboratory tests and animals, IPH2201 has been shown to have effects which result in shrinkage of tumours. IPH2201 has been studied in people with rheumatoid arthritis but it has not yet been studied in people with cancer and the investigators do not know if it can offer better results than standard treatment.

The standard or usual treatment for this disease could include surgery, chemotherapy or radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically and/or cytologically confirmed gynecologic malignancy including high-grade serous ovarian/fallopian tube or peritoneal carcinoma, cervical cancer (squamous cell carcinoma) or endometrial cancer (adenocarcinoma), that is advanced/metastatic/recurrent or unresectable and for which no curative therapy exists.
* For patients with HGSC: For Part 2 of this study, patients will be classified as either platinum resistant or platinum sensitive, as defined by their previous response to platinum-based therapy:

  * The platinum resistant cohort will include patients with disease progression within 6 months of the last line of platinum-based therapy dose.
  * The platinum sensitive cohort will be defined by progression 6 months or longer since last platinum-based therapy dose.
* All patients must have an available formalin fixed paraffin embedded tissue block (from their primary or metastatic tumour) and must have provided informed consent for the release of the block (or slides), as well as for samples for correlative studies and banking.

  • At least 4 patients registered to each cohort in Part 2 must also have provided informed consent for and be willing to undergo a tumour biopsy prior to treatment (after registration) and after treatment with IPH2201. Note: During accrual to Part 2, it may be necessary to restrict accrual to patients who are suitable for, and have consented to, tumour biopsy before and after treatment.
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to randomization/registration (within 35 days if negative).

All patients must have measurable disease as defined by RECIST 1.1. The criteria for defining measurable disease are as follows:

Chest x-ray ≥ 20 mm CT scan (with slice thickness of 5 mm) ≥ 10 mm --> longest diameter Physical exam (using calipers) ≥ 10 mm Lymph nodes by CT scan ≥ 15 mm --> measured in short axis

* Patients must be ≥ 18 years of age.
* Patients must have an ECOG performance status of 0, 1, or 2.
* Previous Therapy
* Cytotoxic Chemotherapy: All patients must have received at least one prior regimen of chemotherapy for advanced, metastatic, or recurrent disease, one of which must have been platinum-based. Patients may have received no more than 3 prior regimens.
* Other systemic therapy: All patients may have received other therapies including immunotherapy, angiogenesis inhibitors, PARP inhibitors or signal transduction inhibitors.
* Patients must have recovered from all reversible toxicity related to prior chemotherapy or systemic therapy and have adequate washout as follows:

Longest of one of the following:

* Two weeks
* 5 half lives for investigational agents
* Standard cycle length of standard therapies

  * Radiation: Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of randomization/registration. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with NCIC CTG.
  * Surgery: Previous surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of randomization/registration, and that wound healing has occurred.

Patients must have recovered from any treatment related toxicities prior to randomization/registration (unless grade 1, irreversible, or considered by investigator as not clinically significant).

* Absolute neutrophils ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 x ULN (upper limit of normal)
* AST and ALT ≤ 2.5 x ULN
* Serum creatinine < 1.25 x ULN ; ≤ 5.0 x UNL if patient has known liver metastases
* Women of childbearing potential must have agreed to use a highly effective contraceptive method during the study and for up to 5 months after the last dose of IPH2201.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to randomization/registration in the trial and prior to tests which are considered to be study specific to document their willingness to participate.
* Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 5 working days of patient randomization (Part 1) or registration (Part 2).

Exclusion Criteria:

* Patients with a history of other active or current malignancies that require active treatment.
* Patients with serious illness or medical conditions that might be aggravated by treatment or limit compliance including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements.
  * Uncontrolled diabetes
  * Active uncontrolled or serious infection (viral, bacterial or fungal)
  * Other medical conditions that might be aggravated by study treatment
* Patients with active immune-mediated diseases or known HIV infection or hepatitis B or C.
* Patients receiving systemic corticosteroid therapy at doses equivalent to more than 5 mg prednisone. Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are permitted.
* Patients receiving cytokines and/or growth factors.
* Patients who have experienced severe adverse effects from other immunotherapy-based treatment or monoclonal antibodies.
* Patients receiving concurrent treatment with other anti-cancer therapy or investigational agents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Dose of single agent IPH2201 for phase II studies and determined based on toxicity, as well as pharmacokinetic and pharmacodynamics data | 24 months
  To confirm the recommended phase II dose (RP2D) of single agent IPH2201 in patients with advanced/metastatic/recurrent platinum sensitive or resistant high-grade serous carcinoma (HGSC) of ovarian, fallopian tube or peritoneal origin.

SECONDARY OUTCOMES:
Number and severity of adverse events in patients | 24 months
  • Safety and tolerability of IPH2201
Correlative assays evaluation for potential predictive markers of IPH2201 effects. Concentration at the end of administration (Cinf end) for all patients | 24 months
  Correlative assays will be used to evaluate potential predictive markers of IPH2201 effects. Other potential prognostic or predictive molecular factors will be assesses in archival tumour tissue, CTCs and blood samples.
Area under the curve from time 0 to Tau=2 weeks (AUC(0-Tau) | 24 months
Accumulation ratio, in terms of Cmax and AUC(0-Tau), between C1 and C4 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hal Hirte, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, ON Canada; Anna Tinker, Study Chair — BCCA - Vancouver Cancer Centre, BC Canada
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tinker AV, Hirte HW, Provencher D, Butler M, Ritter H, Tu D, Azim HA Jr, Paralejas P, Grenier N, Hahn SA, Ramsahai J, Seymour L. Dose-Ranging and Cohort-Expansion Study of Monalizumab (IPH2201) in Patients with Advanced Gynecologic Malignancies: A Trial of the Canadian Cancer Trials Group (CCTG): IND221. Clin Cancer Res. 2019 Oct 15;25(20):6052-6060. doi: 10.1158/1078-0432.CCR-19-0298. Epub 2019 Jul 15. PMID 31308062
- [Derived] Roberto A, Di Vito C, Zaghi E, Mazza EMC, Capucetti A, Calvi M, Tentorio P, Zanon V, Sarina B, Mariotti J, Bramanti S, Tenedini E, Tagliafico E, Bicciato S, Santoro A, Roederer M, Marcenaro E, Castagna L, Lugli E, Mavilio D. The early expansion of anergic NKG2Apos/CD56dim/CD16neg natural killer represents a therapeutic target in haploidentical hematopoietic stem cell transplantation. Haematologica. 2018 Aug;103(8):1390-1402. doi: 10.3324/haematol.2017.186619. Epub 2018 Apr 26. PMID 29700172